CLINICAL TRIAL: NCT02043561
Title: The Effect of Inhibitory Control Processes Induced by Rectal Distension on Impulse Control Measured by Stroop Task Performance and Intertemporal Discounting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: S56275
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2014-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- no urge (Sham Comparator): rectal balloon deflated
  Interventions: Other: induction of urge by rectal distension
- moderate urge (Experimental): moderate urge induced by rectal balloon
  Interventions: Other: induction of urge by rectal distension
- high urge (Experimental): high urge induced by rectal balloon
  Interventions: Other: induction of urge by rectal distension

INTERVENTIONS:
Other: induction of urge by rectal distension

SUMMARY:
The aim of this study will be to investigate the effect of rectal distension, controlled by electronic barostat, on cognitive control ability in healthy subjects. We will use the Stroop task and an intertemporal choice task as standard instruments. Like bladder control and rectal control, both Stroop task performance and intertemporal choices - though very different tasks at the surface - are dependent on the conflict monitoring function of the anterior cingulate cortex. The Stroop task requires the naming of the print color of a series of visually presented color words, and reaction time and error rates are typically used as performance indicators. When word color and word meaning do not match, performance of the task (color naming) requires the inhibition of a (near) automatic response (word reading). The intertemporal choice task consists of a series of choices between a sooner smaller monetary reward and a larger but later reward. The choices are constructed such that they allow the estimation of a discount parameter, which is an index for the level of impulsiveness manifested by the participant at the time the choices are made.

The hypothesis is that the inhibition induced by the urge generated during rectal distension will improve cognitive inhibitory performance, as has previously been shown for bladder filling.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and non-pregnant, non-breastfeeding female participants, aged 18-60 years old at the time of consent.

Exclusion Criteria:

* use of medications within 48 h of dose initiation; structural or metabolic diseases that affect the gastrointestinal system and functional gastrointestinal disorders; previous abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, or hernia repair; known illnesses such as diabetes, cardiovascular or lung disease; current psychiatric disorders (anxiety, depression, substance use); use of agents that influence bowel habit, i.e. anticholinergics (not including antihistamines with anticholinergic properties), spasmolytics and prokinetics in the 7 days before the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2015-09-07 (Actual); Study Completion 2015-09-07 (Actual)

PRIMARY OUTCOMES:
cognitive inhibitory performance on Stroop task (reaction time, in milliseconds) and intertemporal choice task (discount parameter, no unit) | 30 minutes
  * response reaction time on Stroop task
  * discount parameter on intertemporal choice task

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Belgium